CLINICAL TRIAL: NCT01414400
Title: Prospective Study of Bacteremia and Infection Rates Following Cholangioscopy With the Spyglass Cholangioscope
Brief Title: Prospective Study to Investigate the Frequency of Possible Bacterial Entry Into the Bloodstream (Bacteremia) and Infectious Complications Associated With the Use of the Spyglass Cholangioscopy System During ERCP (Endoscopic Retrograde Cholangiopancreatography).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Subhas Banerjee, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-07272011-8148
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Bile Duct Stricture; Choledocholithiasis
Keywords: Bacteremia; Spyglass; Cholangioscopy
MeSH Terms: conditions — Choledocholithiasis; Bacteremia | interventions — Blood Specimen Collection; Culture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Choledochoscopy (Other): Patients undergoing ERCP with choledochoscopy
  Interventions: Other: Blood draw for culture

INTERVENTIONS:
Other: Blood draw for culture — Blood will be drawn and sent for culture.

SUMMARY:
The aim of this study is to prospectively evaluate the frequency of bacteremia after ERCP/cholangioscopy using the Spyglass Direct Visualization System. In addition, the frequency of cholangitis/sepsis despite use of post procedural antibiotics will be studied.

DETAILED DESCRIPTION:
Rates of bacteremia (bacterial seeding of the blood) following ERCP's range from 6.4% to 18.0%. However, infectious complications of cholangitis/sepsis occur in only 0.5%- 3.0% of patients undergoing this procedure. The Spyglass Direct Visualization System allows cholangioscopy with direct visualization of the bile duct during ERCP by using a specialized small caliber endoscope. During the Spyglass portion of the procedure, saline is introduced into the bile duct to to irrigate the biliary system, in order to distend the biliary ducts and to improve visualization by clearing contrast, pus and stone debris. Saline irrigation may increase intrabiliary pressures and may therefore theoretically increase the risk for bacteremia and infection.

The effect of Spyglass cholangioscopy and biliary irrigation on the frequency of bacteremia/post cholangioscopy infections is unknown and has not previously been studied.

The aim of this study is to prospectively evaluate the frequency of bacteremia after ERCP/cholangioscopy using the Spyglass system.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. Biliary disease such as large stones necessitating electrohydraulic lithotripsy;
3. Biliary strictures needing tissue acquisition through cholangioscopic directed biopsies
4. Pancreatic-biliary malignancies needing tissue acquisition through cholangioscopic directed biopsies
5. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Age <18, > 80
2. Potentially vulnerable subjects including pregnant women, homeless people, employees and students.
3. Patients who have a clear indication for pre-procedure antibiotics based on current ASGE guidelines
4. Patients who had received antibiotics for any reason within the prior 7 days
5. Patients who had evidence of systemic infection at time of the ERCP
6. Patients in whom additional venous access for blood cultures cannot be established.
7. Participation in another investigational study within the previous 90 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhas Banerjee, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Thosani N, Zubarik RS, Kochar R, Kothari S, Sardana N, Nguyen T, Banerjee S. Prospective evaluation of bacteremia rates and infectious complications among patients undergoing single-operator choledochoscopy during ERCP. Endoscopy. 2016 May;48(5):424-31. doi: 10.1055/s-0042-101407. Epub 2016 Feb 26. PMID 26919263

RESULTS

PARTICIPANT FLOW:
Groups:
- Choledochoscopy: Patients undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) with choledochoscopy
  Blood draw for culture: Blood drawn and sent for culture.
Period: Overall Study
Arm/Group | Choledochoscopy
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Choledochoscopy
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Bacteremia
Description: This outcome is to assess bacteremia and infection rates in patients following Cholangioscopy with the Spyglass cholangioscope. Positive blood cultures were evaluated for transient ERCP-related bacteremia, and sustained Cholangioscopy-related bacteremia, defined by negative first and second sets of blood cultures but a positive third blood culture obtained 15 minutes after completion of Cholangioscopy and ERCP.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Choledochoscopy: Patients undergoing ERCP with choledochoscopy
  Blood draw for culture: Blood drawn and sent for culture.
Arm/Group | Choledochoscopy
Number analyzed (Participants) | 72
Participants
  Had positive blood culture | 25
  Had true positive blood culture after ERCP/SOC | 20
  Had false positive blood culture due to contaminants | 5
  Had bacteremia following cholangioscopy | 10
  Had bacteremia following ERCP alone | 10
  Had sustained bacteremia following ERCP/Cholangioscopy | 14

ADVERSE EVENTS:
Time Frame: Up to 2 months
Arm/Group | Choledochoscopy
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 20/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Choledochoscopy (N=72)
Bacteremia (Infections and infestations) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No